CLINICAL TRIAL: NCT01028287
Title: "Safety and Efficacy of Acthar Gel on Albuminuria and Urinary Transforming Growth Factor Excretion in Type I or Type II Diabetics Requiring Medical Treatment of Hyperglycemia With Nephrotic Range Proteinuria: A Pilot Study"
Brief Title: Adrenocorticotropic Hormone (ACTH) Treatment of Nephrotic Range Proteinuria in Diabetic Nephropathy (NRDN)
Acronym: ACTH-NRDN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast Renal Research Institute (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, James A. Tumlin MD, Principal Investigator, Southeast Renal Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTH-NRDN
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Nephropathy; Nephrotic Syndrome
Keywords: Diabetic Nephropathy; Nephrotic syndrome
MeSH Terms: conditions — Diabetic Nephropathies; Nephrotic Syndrome | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTH-16 units (Active Comparator): Patients with nephrotic range proteinuria randomized to this group will receive 16 units ACTHargel sub-cutaneously every day.
  Interventions: Drug: ACTH
- ACTH-32 units (Active Comparator): Patients with nephrotic range proteinuria randomized to this group will receive 32 units ACTHargel sub-cutaneously every day.
  Interventions: Drug: ACTH

INTERVENTIONS:
Drug: ACTH — Patients with nephrotic range proteinuria randomized to this group will receive 16 units ACTHargel sub-cutaneously every day.
  Other Names: ACTHar Gel
Drug: ACTH — Patients with nephrotic range proteinuria randomized to this group will receive 32 units ACTHargel sub-cutaneously every day.
  Other Names: ACTHar Gel

SUMMARY:
This is a prospective open labeled trial examining the efficacy of ACTHar Gel (porcine ACTH) on the level of proteinuria in patients with diabetic nephropathy and nephrotic range proteinuria.

DETAILED DESCRIPTION:
Diabetes Mellitus is a significant and growing health problem in the United States and other developed countries. Despite improving public awareness, end-organ complications including diabetic nephropathy and coronary atherosclerotic heart disease continues to grow by 5-10% per year. While improvements in the control of blood pressure and the wide-spread use of antagonists of the renin-angiotensin-aldosterone system have significantly improved renal outcomes, therapies designed to disrupt the more central pathogenic mechanisms of diabetic nephropathy are still needed. Recent observations have shown that effacement of podocyte foot-plate processes and accelerated apoptosis, are central to the pathogenesis of diabetic nephropathy. The resulting increase in glomerular permeability leads to nephrotic range proteinuria and interstitial fibrosis from local synthesis of transforming growth factor b (TGF-b) and direct toxicity to the renal epithelium. Recent studies have shown that synthetic forms of adrenocorticotropic hormone (ACTH) are able to achieve sustained reductions in proteinuria in non-diabetic glomerulopathies. Moreover, while the numbers of patients are quite limited, preliminary studies also suggest that pharmacologic administration of ACTH can reduce proteinuria in patients with diabetic nephropathy. The observation that ACTH can reduce proteinuria in a variety of glomerulopathies suggests that ACTH may be important for podocyte function and viability independent of the primary disease. Interestingly, recent studies confirm that melanocortin receptors are expressed in non-adrenal tissues including the circulating T and B cells and most recently the glomerular podocyte. Previous studies investigating the effect of diabetes and insulin therapy on ACTH levels have given mixed results. It is therefore unclear how podocytes in patients with diabetic nephropathy could become functionally deficient in ACTH. However, studies in adrenal cortical cells finds that TGF-b is able to down regulate the expression of ACTH receptors. Moreover, TGF-b is able block an ACTH-induced stimulation of melanocortin receptors. This intriguing link between TGF-b and ACTH signaling raises the question of whether impaired signaling of ACTH in the glomerulus leads to podocyte dysfunction, accelerated detachment and ultimately podocyte apoptosis. Moreover, we postulate that a complex interaction between TGF-b and ACTH expression exists within the glomerulus such that restoration of ACTH function will lead to a reduction in renal TGF-b expression. We therefore propose to study the effect of increasing doses of exogenous ACTH on rates of albuminuria and urinary TGF-b expression in diabetics with nephrotic range proteinuria. In addition to TGF-b we will examine whether a similar effect occurs on the 3 major isoforms of vascular endothelial growth factor, VEGF120, 164, and 180. We will also determine the duration of the effect and whether it is additive with ACE/ARB therapy inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 80
2. Type I or Type II Diabetes Mellitus
3. Stable ACE or ARB therapy for 4 weeks prior to study enrollment
4. Urinary protein > 3000 mg/24 hrs
5. Patients with more than one protein lowering agent (e.g. ACE or ARB, or MR antagonist or Tekturna require two consecutive 24 hour urinary protein of 2000 mg/24 hrs.

Exclusion Criteria:

1. Age <18 or >80
2. HgbA1c > 9.0% or 11% if using the (DCCT / NGSP) method.
3. eGFR < 20 mls/min by MDRD formula or eGFR by (Cockoff-Gault 20 mls/min)
4. Dilated cardiomyopathy with known EF < 40%
5. Pregnant or nursing mothers
6. Patients with an admission for diabetic ketoacidosis, or non-ketotic hyperosmolar coma within 6 months of study enrollment.
7. Patients with known mixed glomerulonephritis and diabetic glomerulopathy
8. Patients within 3 mths of operative procedures or chronic non-healing wounds
9. Patients with glucocorticoid-induced diabetes mellitus
10. Patients with known sensitivity to porcine protein products
11. Patients with bleeding gastric or duodenal ulcers requiring hospitalization six months prior to study enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving less than 300 mg protein per 24 hours after 6 months of Acthar Gel. | 6 months

SECONDARY OUTCOMES:
Percentage of patients achieving greater than 50% reduction in urinary proteinuria after 6 months of Acthar Gel. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tumlin, MD, Principal Investigator — Southeast Renal Research Institute
Locations (1):
- Southeast Renal Research Institute, Chattanooga, Tennessee, United States

REFERENCES:
- [Derived] Tumlin JA, Galphin CM, Rovin BH. Advanced diabetic nephropathy with nephrotic range proteinuria: a pilot study of the long-term efficacy of subcutaneous ACTH gel on proteinuria, progression of CKD, and urinary levels of VEGF and MCP-1. J Diabetes Res. 2013;2013:489869. doi: 10.1155/2013/489869. Epub 2013 Sep 12. PMID 24159603